CLINICAL TRIAL: NCT07035808
Title: Efficacy and Safety of Iparomlimab and Tuvonralimab(QL1706) Combined With Chemotherapy ± Bevacizumab Induction Therapy Followed by Concurrent Chemoradiotherapy for High-risk Locally Advanced Cervical Cancer：a Single Arm, Phase II Multicenter Clinical Study
Brief Title: a Single Arm, Phase II Multicenter Clinical Trial to Evaluate the Efficacy and Safety of the Combination Therapy of Iparomlimab and Tuvonralima b and Chemotherapy ± Bevacizumab Induction Therapy Followed by Concurrent Chemoradiotherapy in Patients With Advanced Cervical Cancer .
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Cancer Hospital of The University of Chinese Academy of Sciences (Unknown); Cancer Center of the First Affiliated Hospital of Soochow University (Unknown); The First Affiliated Hospital of Nanchang University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); People's Hospital of Quzhou (Other); First Affiliated Hospital of Ningbo University (Network); Wenzhou Central Hospital (Other); Jinhua Municipal Central Hospital (Other); First Hospital of Zhejiang University (Unknown); First Affiliated Hospital of Zhejiang University (Other); Henan Provincial People's Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hanmei Lou, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-2025-086
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer Stage IVA; Cervical Cancer Metastatic
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Combination Product: 2 cycles of combined drug induction therapy: every 3 weeks for 2 cycles; After ,synchronous radiotherapy and chemotherapy combined immunotherapy

INTERVENTIONS:
Combination Product: 2 cycles of combined drug induction therapy: every 3 weeks for 2 cycles; After ,synchronous radiotherapy and chemotherapy combined immunotherapy — The enrolled patients first receive 2 cycles of combined drug induction therapy: paclitaxel+cisplatin/carboplatin ± bevacizumab+QL1706, every 3 weeks for 2 cycles; After induction therapy, synchronous radiotherapy and chemotherapy combined with immunotherapy: extracorporeal irradiation+post loading radiotherapy+synchronous chemotherapy+immunotherapy. During radiotherapy, single agent cisplatin/carboplatin treatment for 5 courses per week+QL1706 treatment every 3 weeks for 3 courses; After the end of radiotherapy and chemotherapy, immune maintenance therapy will be administered for six months: treatment with QL1706 every 3 weeks for 9 courses, followed by a follow-up period until the end of radiotherapy for 2 years or death.

SUMMARY:
This study is a single arm, phase II multicenter clinical trial to evaluate the efficacy and safety of the combination therapy of Iparomlimab and Tuvonralimab(QL1706) and chemotherapy ± bevacizumab induction therapy followed by concurrent chemoradiotherapy in patients with locally advanced cervical cancer at high risk of IVA stage and/or giant cervical tumors and/or giant metastatic lymph nodes and/or multiple metastatic lymph nodes.

The enrolled patients first receive 2 cycles of combined drug induction therapy: paclitaxel+cisplatin/carboplatin ± bevacizumab+QL1706, every 3 weeks for 2 cycles; After induction therapy, synchronous radiotherapy and chemotherapy combined with immunotherapy: extracorporeal irradiation+post loading radiotherapy+synchronous chemotherapy+immunotherapy. During radiotherapy, single agent cisplatin/carboplatin treatment for 5 courses per week+QL1706 treatment every 3 weeks for 3 courses; After the end of radiotherapy and chemotherapy, immune maintenance therapy will be administered for six months: treatment with QL1706 every 3 weeks for 9 courses, followed by a follow-up period until the end of radiotherapy for 2 years or death.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign a written informed consent before any trial-related procedures. 2. Histologically confirmed cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma.

  3. Patients with stage Ⅳa confirmed by endoscopic biopsy and/or stage IB3-IIIC (FIGO 2018 staging) with large cervical tumors (maximum diameter ≥ 6 cm) and/or large lymph nodes (maximum short diameter of cross-section ≥ 2 cm) and/or ≥ 3 lymph node metastases confirmed by CT/MR/PET.

  4. Female patients aged ≥ 18 years and ≤ 75 years. 5. KPS ≥ 70. 6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

  7. Expected survival of more than 6 months. 8. No previous radiotherapy, chemotherapy, immunotherapy or targeted therapy. 9. Major organ functions meet the following requirements: Absolute neutrophil count ≥ 1.5×109/L, platelet count ≥ 80×109/L, hemoglobin ≥ 80g/L; Total bilirubin level ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN; Serum creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 60 ml/min; Serum albumin ≥ 28g/L; thyroid stimulating hormone (TSH) ≤ 1×ULN (if abnormal, FT3 and FT4 levels should also be examined. If FT3 and FT4 levels are normal, the subject can be enrolled).

  10. Subjects agree to use effective contraceptive measures from the time of signing the informed consent until 180 days after the last dose. Women of childbearing age must not be pregnant or lactating.

  11. All subjects must be willing to provide tumor tissue samples, blood samples, urine samples, fecal samples, and vaginal secretion samples after enrollment.

Exclusion Criteria:

1. Other histopathological findings such as neuroendocrine carcinoma, sarcoma, gastric-type adenocarcinoma, and malignant melanoma components;
2. Previous receipt of anti-tumor treatment related to cervical cancer;
3. Evidence of distant metastasis, including lymph node metastasis in the groin, supraclavicular, and axillary regions;
4. Previous total hysterectomy or subtotal hysterectomy;
5. Anatomical abnormalities or contraindications that preclude the use of brachytherapy;
6. Previous receipt of any treatment targeting tumor immune mechanisms, such as immune checkpoint inhibitors (e.g., anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies) or antibodies targeting immune co-stimulatory factors (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40 targets);
7. Patients with other tumors that require current treatment;
8. Active or potentially recurrent autoimmune diseases, except for those that do not require systemic treatment: vitiligo, alopecia, psoriasis or eczema; hypothyroidism caused by autoimmune thyroiditis, requiring stable doses of hormone replacement therapy; type 1 diabetes requiring stable doses of insulin replacement therapy;
9. Patients currently using immunosuppressants or systemic hormones to achieve immunosuppression, and still using them within 2 weeks before enrollment;
10. Poorly controlled clinical symptoms or diseases of the heart, such as (1) NYHA grade 2 or above heart failure; (2) unstable angina pectoris; (3) severe myocardial infarction within 1 year; (4) need for treatment or intervention for clinically significant supraventricular or ventricular arrhythmias; (5) QTc > 450 ms (male), QTc > 470 ms (female);
11. Abnormal coagulation function (INR > 2.0, PT > 16s);
12. Known hereditary or acquired bleeding disorders or thrombophilia (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, etc.);
13. Congenital or acquired immune deficiencies (such as HIV-infected individuals);
14. Patients with HBV DNA > 2000 IU/ml, or HCV RNA > 103, or HBsAg + anti-HCV antibody positive;
15. Active infections that require treatment or use of systemic anti-infective drugs within one week before the first administration;
16. Within 4 weeks before the first administration, received major surgical treatment or had significant trauma or required elective major surgical treatment during the study period.
17. Hypertension, and unable to achieve good control with antihypertensive drugs (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg); previous occurrence of hypertensive crisis or hypertensive encephalopathy;
18. Known that the patient was previously allergic to large molecule protein preparations. Has contraindications and allergies to epalorlimovalovirumab, cisplatin, carboplatin, paclitaxel, bevacizumab, any components thereof;
19. Presence of abnormal results that may interfere with the test results, prevent the subject from fully participating in the study, or laboratory abnormalities that the investigator considers not in the best interests of the subject.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year PFS | 2 year
  2-year PFS rate evaluated by researchers based on RECIST v1.1 and biopsy pathology

SECONDARY OUTCOMES:
ORR | 2 year
  ORR of drug-induced therapy evaluated by researchers based on RECIST v1.1 and biopsy pathology
DCR | 2 year
  DCR of drug-induced therapy evaluated by researchers based on RECIST v1.1 and biopsy pathology
OS | 2 year
  2-year OS

IPD SHARING:
Plan to Share IPD: No